CLINICAL TRIAL: NCT00598065
Title: The Use of Breathing Synchronized PET/CT Imaging In the Detection and Quantification of FDG Uptake in Lung Nodules
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Memorial Sloan Kettering Cancer Center (Other)
Responsible Party: Schoder, Heiko, MD / Principal Investigator, Memorial Sloan-Kettering Cancer Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 04-025
Record Dates: First submitted 2008-01-09; First posted 2008-01-18 (Estimated); Last update posted 2009-12-03 (Estimated); Status verified 2009-12

CONDITIONS: Lung Cancer
Keywords: lung
MeSH Terms: conditions — Lung Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Other: PET/CT — Synchronized PET/CT Imaging

SUMMARY:
The purpose of this study is to see if researchers can improve the detection of lung cancer by using a new method which will help us to take multiple snapshot images of the lungs while the patient is breathing. We are also investigating whether with the help of this new method we can better measure the actual amount of radioactivity that is taken up by the cancer. The name of this new method is respiratory gated PET/CT. Previous research has shown that PET scans may be useful in investigating whether cancer has spread to other parts of the lung or body. Using our standard method, smaller cancers are sometimes difficult to detect in the lungs because the PET images are taken over several minutes and the patient is breathing during that time. That means the cancer may appear "blurred" on the images (like a poor photograph) or may not be identified at all. In this study, in addition to the images that were ordered by your doctor, we will take additional images of your lungs while you are following a breathing command ("breath in-hold-breath out"). We will then compare the images of your cancer during the regular PET study with those taken during the breathing commands.

The hypotheses to be tested in this pilot study are:

1. Respiratory gated image acquisition reduces partial volume effects on PET image that may render lung lesions undetectable.
2. Breath-hold CT may detect small lung lesions that are beyond the limit of detection in shallow-breathing CT scans, related to respiratory motion which causes blurring artifacts around smaller lung lesions.

DETAILED DESCRIPTION:
Positron emission tomography is now a clinically accepted imaging modality for the evaluation of pulmonary nodules as well as for the staging of patients with lung cancer. PET imaging with the radiotracer 18 Fluoro-deoxy-glucose (FDG) has a high accuracy for the differentiation between benign and malignant lung lesions and for the detection of nodal metastases. This is because malignant tumors are characterized by an increase in glucose metabolism as compared to most normal tissues. In clinical practice, PET images are interpreted visually or semiquantitatively, using a standardized uptake value (SUV). Previous studies have shown that SUV thresholds can be used with high accuracy to distinguish between benign and malignant lesions that exhibit increased uptake of FDG. In addition, the SUV is frequently used as a surrogate marker for the evaluation of a response to chemo- or radiation therapy. Unfortunately, the accuracy of SUV measurements may be affected by lesion motion during the image acquisition. This is a particular problem in PET imaging of the lung. Normal respiratory motion, and hence lesion motion, causes a smearing effect, whereby the concentration of radiotracer within a given lesion is spread out over a larger area. For the same reason small lesions and lesions with relatively low uptake of radiotracer may become undetectable during normal breathing (partial volume effect). PET images are acquired for several minutes, image acquisition during breath hold is therefore not an option for clinical scans. However recently published work from UCLA (Auerbach et al. J Nucl Med., February 2006) shows that 3 lesions per patient on average can be missed on shallow breathing scans compared to breath-hold CT scans. These lesions did not show any FDG uptake on clinical PET scans. The goal of this pilot study is to evaluate whether respiratory gating during PET image acquisition enables the detection of those lesions which are identified during the breath-hold CT scan.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years old
* Patients must have at least one lung lesion or lung cancer on prior chest Xray or chest CT.
* Sign informed consent. Eligible patients should give their consent at the beginning of the clinical PET scan. Following clinical CT and PET scans, breathhold CT should follow. Then, these breath-hold CT images will be reviewed by one of the investigating physicians to determine if the patient qualifies for the study. If there is a small lesion (< 5 mm) gated PET images will be acquired.

Exclusion Criteria:

* Pregnant women are ineligible.
* Patients who are unable to follow breathing instructions either due to language difficulties or hearing impairment This will be determined by one of the consenting individuals when they approach the patient to ask for informed consent.
* Patients who are too ill to hold their breath.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 26 (Actual)
Dates: Start 2004-03; Primary Completion 2009-12 (Actual); Study Completion 2009-12 (Actual)

PRIMARY OUTCOMES:
Pts w/suspected lung lesions will undergo more breath-hold CT scan & if visible lesion(s), gated-PET will be acquired plus clinical PET/CT. Scans will be used to compare how often additional lung lesions can be identified on breath-hold CT, if lesions | 5 years

CONTACTS AND LOCATIONS:
Overall Officials: Heiko Schoder, MD, Principal Investigator — Memorial Sloan Kettering Cancer Center
Locations (1):
- Memorial Sloan Kettering Cancer Center, New York, New York, United States

REFERENCES:
- See also: Memorial Sloan-Kettering Cancer Center — http://www.mskcc.org